CLINICAL TRIAL: NCT05785078
Title: Evaluation of the Impact of a Program to Raise Awareness About Flu Vaccination and a Vaccination Campaign Aimed at Women Participating in the Childbirth Preparation Course Held at Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Brief Title: Evaluation of a Flu Vaccination Program Directed at Pregnant Women Assisted at a Research Hospital in Italy.
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2782
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Educational session about vaccinations — An educational session about maternal and childhood vaccinations was held in the context of the Childbirth Preparation Course held monthly at the FPG. In this occasion, on-site flu vaccination was offered to pregnant women attending the course and their partners, if present.

SUMMARY:
Influenza is a serious Public Health problem, which causes a high number of cases and deaths worldwide each year. In Italy, about 8 million cases were reported in the 2018/2019 flu season, 809 of which were severe, with 198 deaths. Pregnant women are considered one of the most at-risk groups, as infection can lead to serious complications for the mother and fetus. The Italian Ministry of Health recommends free flu vaccination for pregnant women in the second or third trimester, as the vaccine is safe and effective in protecting the mother, fetus and newborn.

During the 2018-2019 flu season, the Fondazione Policlinico Universitario A. Gemelli IRCCS (FPG) held an educational session on maternal and childhood vaccinations in the context of the Childbirth Preparation Course held monthly at the FPG, offering the on-site flu vaccination to participants and their partners, if present.

The objectives of this study are: to improve knowledge and attitudes regarding vaccination in the course participants, assessing their changes through a pre-post anonymous questionnaire; to evaluate the impact of the flu vaccination strategy implemented, through the analysis of vaccination coverage.

ELIGIBILITY:
Inclusion Criteria:

* Attendance to the educational session about vaccination in the context of the childbirth preparatory course held at Fondazione Policlinico Universitario "A. Gemelli" IRRCS

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women and their partners attending the childbirth preparatory course held at Fondazione Policlinico Universitario "A. Gemelli" IRRCS
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Differences in knowledge and attitudes regarding vaccination | 4 months
  Change in Knowledge and Attitudes About Vaccination from Pre- to Post-Educational Session

SECONDARY OUTCOMES:
Vaccination compliance | 4 months
  Number of Participants Compliant with On-site Influenza Vaccination Offer

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No